CLINICAL TRIAL: NCT07246395
Title: Narrative Family Therapy in Autism Spectrum: From Clinical Neuroscience to Intervention Outcomes
Brief Title: NarraTivAS - Narrative Family Therapy in Autism Spectrum
Acronym: NarraTivAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Miguel Castelo-Branco, Full Professor, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NarraTivASD01CIBIT; 2021.05559.BD (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia (FCT)); UID/4950/2025 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia (FCT))
Record Dates: First submitted 2025-09-11; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Narrative Family Therapy; Family Functioning; Therapeutic Change
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): The control group will receive a family-based intervention grounded in Game Theory.
  Interventions: Behavioral: Family Game Theory-based Intervention
- Experimental Arm (Experimental): The experimental group will receive Narrative Family Therapy for Autism Spectrum Disorder, a brief manualized intervention.
  Interventions: Behavioral: Narrative Family Therapy

INTERVENTIONS:
Behavioral: Narrative Family Therapy — Participants in the intervention group will attend eight Narrative Family Therapy sessions, each lasting 60-90 minutes with one therapist. The first four sessions occur weekly; the remaining are monthly, with a follow-up three months after the final session. This brief, manualized therapy was developed to address the specific needs of families with autistic members. It uses sensory materials and preferred topics as entry points for therapeutic dialogue. Each session begins with the autistic individual and concludes by asking each participant to share what they took from the session. Information is presented visually (e.g., brain style profile) to match the visual strengths of individuals with autism. The intervention aims to promote narrative transformation, leading to changes in stories, relationships, and perspectives. These shifts help participants express and organize their experiences more adaptively, supporting improved interpersonal relationships and functioning.
  Arms: Experimental Arm
Behavioral: Family Game Theory-based Intervention — The control group will receive a Family Game Theory-based approach consisting of eight sessions, each lasting 60-90 minutes and conducted without a therapist. The first four sessions are held weekly, while the remaining sessions occur monthly, followed by a final follow-up three months after the last session. This approach was designed to reflect family dynamics through three classical game theory models: the Stag Hunt, the Prisoner´s Dilemma, and the Battle of the Sexes. Each session begins with a phase in which family members are invited to share something with one another. Then, they participate in a round of non-verbal dyadic games using a tablet. Finally, they are encouraged to reflect and share what they took from the session.
  Arms: Control Arm

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopmental condition characterized by difficulties in social communication and interaction, along with restricted and repetitive patterns of behavior, interests, or activities. While previous research has largely focused on individualized therapies and behavioral outcomes for people with autism, there remains a gap in understanding the broader effect on family systems functioning and the neurobiological changes that may occur following intervention.

This project aims to address that gap by characterizing families of individuals with autism, examining both individual and family-level variables, including their motivation to participate in Narrative Family Therapy. Participating families will be assigned to either an intervention group receiving Narrative Family Therapy or a control group engaged in a Game Theory-based approach (e.g., Stag Hunt Dilemma, Prisoner's Dilemma, War of the Sexes), designed to reflect family dynamics.

A mixed-methods approach will be employed to explore therapeutic changes across three key areas: (1) theory-of-mind brain networks, (2) narrative change, and (3) the overall well-being of family members reflected by the family functioning perceptions. Neurobiological data will be collected via functional Magnetic Resonance Imaging (fMRI) during an autobiographical, therapy-related task, conducted both before and after the intervention. This will be complemented by physiological measurements-including galvanic skin response (GSR), respiratory sinus arrhythmia (RSA), and heart rate variability (HRV)-to evaluate autonomic nervous system activity.

The investigators hypothesize that Narrative Family Therapy may promote neuroplasticity and restore effective connectivity within core brain circuits associated with social cognition, particularly the amygdala, ventromedial prefrontal cortex, and temporoparietal junction. Physiological data (GSR, HRV) collected during therapy sessions will also be analyzed to measure session-level effects. Specifically, the investigators will test whether autonomic arousal decreases across sessions and whether this reduction correlates with narrative development, assessed using the Assessment System of Narrative Change (ASNC) - a qualitative method based on empirical findings in Narrative Family Therapy.

To assess the feasibility and effectiveness of the therapeutic protocol, the Systemic Clinical Outcome and Routine Evaluation Scale (SCORE-15) and the Family Adaptability Cohesion Evaluation Scales IV Version (FACES-IV) will be administered. The investigators expect that the intervention will reduce mental health issues and enhance family functioning-such as communication, flexibility, and satisfaction-compared to the control group.

Overall, this study seeks to advance both scientific knowledge and clinical practice by fostering an innovative dialogue between Narrative Family Therapy and neuroscience.

ELIGIBILITY:
Inclusion Criteria:

* Families of children, adolescents and/or young adults with ages ranging from 8 to 18 years;
* Children, adolescents and/or young adults with a primary diagnosis of Autism Spectrum Disorder, verbally fluent, and without intellectual impairment (intelligence quotient above 70 as measured by the Wechsler Intelligence Scale for Children or Adults - 3rd Edition, WISC-III or WAIS-III).
* Nuclear intact, divorced, large, and single-parent families.

Exclusion Criteria:

* Participants with brain injury, alcoholism, drug abuse, active psychosis, homicidal/suicidal ideation, and personality disorder.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to the post-intervention in the Systemic Clinical Outcome Routine Evaluation - 15 items (SCORE-15) | From baseline to the end of treatment at 5 months.

SECONDARY OUTCOMES:
Change from baseline to the post-intervention (5 months) and follow up (8 months later) in the Portuguese Family Communication and Family Cohesion - Version IV | From baseline to the end of treatment at 5 months, and to follow-up to 8 months (from baseline).
Assessment System of Narrative Change | At each intervention session from first to last (intervention last 5 months) and at follow-up (after 3 months from the last intervention session).
  A coding system will assess the narrative change - the Assessment System of Narrative Change (Sequeira & Alarcão, 2013). This system was developed to assess and classify narratives expressed in therapy to trace changes over the course of therapy (Sequeira & Alarcão, 2013). The coding measure that will be used will cover areas of narrative change such as: Total number of specific codes in each session (please cf. Sequeira & Alarcão, 2013). The measure will be used to code transcripts on a session-by-session basis and is therefore a process measure.
BOLD changes from baseline to the post intervention (5 months) | Assessments will be conducted within two weeks prior to the first intervention session and within two weeks following the end of the intervention (at five months).
  BOLD signal changes from baseline to the post intervention (5 months), during an Functional Magnetic Imaging Ressonance (fMRI) task of visualization of autobiographical images
The Satisfaction with Therapy and Therapist Scale-Revised adaptation after the follow-up (8 months) | After the follow-up session (8 months from baseline) within a month.
The long-term effect from pre-baseline (before intervention study enrollment) to the follow-up session on the Social Responsivness Scale- 16 items scores. | From pre-baseline (before the enrolment on the intervention study) to follow up within a month after the follow-up.
The long-term effect from pre-baseline (before intervention study enrollment) to the follow-up session on Brief Measure of Parental Wellbeing | From pre-baseline (before the enrolment on the intervention study) to follow up within a month after the follow-up.
The long-term effect from pre-baseline (before intervention study enrollment) to the follow-up session on Walsh Family Resilience Questionnaire | From pre-baseline (before the enrolment on the intervention study) to follow up within a month after the follow-up.
The long-term effect from pre-baseline (before intervention study enrollment) to the follow-up session on Coparenting Questionnaire | From pre-baseline (before the enrolment on the intervention study) to follow up within a month after the follow-up.
Skin Conductance Response | At each intervention session from first to last (intervention last 5 months) and at follow-up (after 3 months from the last intervention session

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Nuclear Sciences Applied to Health (ICNAS), University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided